CLINICAL TRIAL: NCT05536726
Title: A Phase 3, Multicenter, Randomized, Double-blind, Placebo-controlled Trial to Evaluate the Efficacy and Safety of Recombinant Anti-IL-17A Humanized Monoclonal Antibody in Chinese Patients With Moderate-to-Severe Plaque Psoriasis
Brief Title: A Phase 3 Study of Recombinant Anti-IL-17A Humanized Monoclonal Antibody in Chinese Participants With Moderate-to-Severe Plaque Psoriasis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sunshine Guojian Pharmaceutical (Shanghai) Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SSGJ-608-PsO-III-01
Record Dates: First submitted 2022-09-08; First posted 2022-09-13 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: Psoriasis
MeSH Terms: conditions — Psoriasis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- 608 160 mg W0+80 mg Q2W+80 mg Q4W (Experimental): Participants will receive starting dose of 160 milligrams (mg) 608 at week 0 followed by 80mg 608 once every two weeks (Q2W) by subcutaneous injection during induction period (12 weeks). During the maintenance period, participants will receive 80mg 608 once every four weeks (Q4W).
  Interventions: Drug: 608 Q2W
- 608 160 mg Q4W+160 mg Q8W (Experimental): Participants will receive 160mg 608 once every four weeks (Q4W) by subcutaneous injection during induction period (12 weeks) followed by 160mg 608 once every eight weeks (Q8W) during maintenance period.
  Interventions: Drug: 608 Q4W
- Placebo (Placebo Comparator): Participants will receive Placebo by subcutaneous injection during induction period and then, will be re-randomized to either receive starting dose of 160mg 608 at week 12 followed by 80mg 608 once every four weeks (Q4W) or 160mg 608 once every eight weeks (Q8W) during maintenance period.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: 608 Q2W — 608 160 mg at week 0 + 80 mg Q2W ( 6 cycles) +80 mg Q4W during maintenance period
  Arms: 608 160 mg W0+80 mg Q2W+80 mg Q4W
Drug: 608 Q4W — 608 160 mg Q4W ( 3 cycles) +160 mg Q8W during maintenance period
  Arms: 608 160 mg Q4W+160 mg Q8W
Drug: Placebo — Participants will receive Placebo at pre-specified time points to maintain the blinding of the Investigational Medicinal Products.
  Other Names: PBO
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine the efficacy and safety of the study drug recombinant anti-IL-17A humanized monoclonal antibody in Chinese participants with moderate-to-severe plaque psoriasis.

DETAILED DESCRIPTION:
Study SSGJ-608-PsO-III-01 is a phase 3, multicenter, randomized, double-blind, placebo-controlled, parallel-group study examining the effect of 2 dose regimens of recombinant anti-IL-17A humanized monoclonal antibody versus placebo in Chinese participants with moderate-to-severe plaque psoriasis during an induction dosing period with dosing for 12 weeks and the primary endpoint measured at 12 weeks, followed by a randomized, double-blind, 40-week maintenance dosing period. During the maintenance dosing period, the study will evaluate the maintenance of response/remission, as well as relapse following treatment.

ELIGIBILITY:
Inclusion Criteria:

* Must be 18 Years to 75 Years, both male and female.
* Chronic plaque psoriasis (PSO) for at least 6 months prior to the Randomization.
* Psoriasis Area Severity Index (PASI) >=12 and body surface area (BSA) affected by PSO >=10% and Static Physician Global Assessment (sPGA) score >=3.
* According to the judgment of the investigator, the subject needs to receive systemic treatment and / or phototherapy (including subjects who have used local treatment, and / or phototherapy, and / or poor control of previous systemic treatment).
* Fertile female subjects and male subjects (and their female partners) must take effective contraceptive measures within at least 6 months from the screening period to the last medication. The subjects have no fertility, sperm donation and egg donation plans within at least 6 months from the screening period to the last medication.

Exclusion Criteria:

* Forms of psoriasis other than chronic plaque-type (e.g., pustular, erythrodermic and/or guttate psoriasis) at screening or baseline.
* Drug-induced psoriasis.
* Ongoing use of prohibited treatments.
* Have previously received any drug that directly targets IL-17 or IL-17 receptor, or IL-12 / IL-23, or IL-23.
* Biological agents or their biological analogues were used before randomization, including but not limited to: Etanercept < 28 days; Infliximab, adalimumab or afacet <60 days; Golimumab <90 days; Or other biological agents < 5 half lives.
* Pregnant or lactating women.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 458 (Actual)
Dates: Start 2023-01-07 (Actual); Primary Completion 2023-10-20 (Actual); Study Completion 2024-06-04 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants Achieving a ≥75% Improvement in Psoriasis Area and Severity Index (PASI 75) | At Week 12
  The PASI combines the extent of body surface involvement in 4 anatomical regions (head, trunk, arms, and legs). For each region the percent area of skin involved was estimated from 0 (0%) to 6 (90%-100%) and severity was estimated by clinical signs of erythema, induration and scaling with a scores range from 0 (no involvement) to 4 (severe involvement). Each area is scored by itself and the scores then combined for the final PASI. Final PASI calculated as: sum of severity parameters for each region * area score * weighing factor [head (0.1), upper limbs (0.2), trunk (0.3), lower limbs(0.4)]. Overall scores range from 0 (no Ps) to 72 (the most severe disease).
Percentage of Participants With a Static Physician Global Assessment (sPGA) Score of Clear (0) or Minimal (1) With at Least a 2 Point Improvement | At Week 12
  The sPGA is the physician's determination of the participant's Ps lesions overall at a given time point. Lesions were categorized by descriptions for induration, erythema, and scaling. Participants Ps were assessed as 0 (clear), 1 (minimal), 2 (mild), 3 (moderate), 4 (severe), or 5 (very severe). An sPGA responder was defined as having a postbaseline sPGA score of "0" or "1" with at least a 2-point improvement from baseline.

SECONDARY OUTCOMES:
Key Secondary: Percentage of Participants Achieving a ≥90% Improvement in Psoriasis Area and Severity Index (PASI 90) | At Week 12
  The PASI combines the extent of body surface involvement in 4 anatomical regions (head, trunk, arms, and legs). For each region the percent area of skin involved was estimated from 0 (0%) to 6 (90%-100%) and severity was estimated by clinical signs of erythema, induration and scaling with a scores range from 0 (no involvement) to 4 (severe involvement). Each area is scored by itself and the scores then combined for the final PASI. Final PASI calculated as: sum of severity parameters for each region * area score * weighing factor [head (0.1), upper limbs (0.2), trunk (0.3), lower limbs(0.4)]. Overall scores range from 0 (no Ps) to 72 (the most severe disease).
Key Secondary: Percentage of Participants Achieving a 100% Improvement in Psoriasis Area and Severity Index (PASI 100) | At Week 12
  The PASI combines the extent of body surface involvement in 4 anatomical regions (head, trunk, arms, and legs). For each region the percent area of skin involved was estimated from 0 (0%) to 6 (90%-100%) and severity was estimated by clinical signs of erythema, induration and scaling with a scores range from 0 (no involvement) to 4 (severe involvement). Each area is scored by itself and the scores then combined for the final PASI. Final PASI calculated as: sum of severity parameters for each region * area score * weighing factor [head (0.1), upper limbs (0.2), trunk (0.3), lower limbs(0.4)]. Overall scores range from 0 (no Ps) to 72 (the most severe disease).
Key Secondary: Percentage of Participants Achieving a Static Physician Global Assessment (sPGA) Score of Clear (0) | At Week 12
  The sPGA is the physician's determination of the participant's Ps lesions overall at a given time point. Lesions were categorized by descriptions for induration, erythema, and scaling. Participants Ps were assessed as 0 (clear), 1 (minimal), 2 (mild), 3 (moderate), 4 (severe), or 5 (very severe).
In the IMP Group, Percentage of Participants Still Maintaining PASI 75, PASI 90 and sPGA 0/1 At Week 52 From Week 12 for Participants Who Achieved PASI 75, PASI 90 and sPGA 0/1 | At Week 52
  The PASI combines the extent of body surface involvement in 4 anatomical regions (head, trunk, arms, and legs). For each region the percent area of skin involved was estimated from 0 (0%) to 6 (90%100%) and severity was estimated by clinical signs of erythema, induration and scaling with a scores range from 0 (no involvement) to 4 (severe involvement). Each area is scored by itself and the scores then combined for the final PASI. Final PASI calculated as: sum of severity parameters for each region * area score * weighing factor [head (0.1), upper limbs (0.2), trunk (0.3), lower limbs(0.4)]. Overall scores range from 0 (no Ps) to 72 (the most severe disease).
Percentage of Participants Achieving an Itch Numeric Rating Scale (NRS) ≥4 Point Reduction From Baseline for Participants Who Had Baseline Itch NRS ≥4 | At Week 12
  The Itch NRS is a participant-administered, 11-point horizontal scale anchored at 0 (no itch) and 10 (worst itch imaginable). Overall severity of a participant's itching from Ps is indicated by circling the number that best describes the worst level of itching in the past 24 hours.

CONTACTS AND LOCATIONS:
Overall Officials: Jinhua Xu, MD, Principal Investigator — Shanghai Huanshan Hospital Fudan University-Dermatology; Jing Zhang, MD, Principal Investigator — Shanghai Huanshan Hospital Fudan University; Qinghong Zhou, MD, Study Director — Sunshine Guojian Pharmaceutical (Shanghai) Co., Ltd.
Locations (1):
- Shanghai Huanshan Hospital Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No